CLINICAL TRIAL: NCT04298853
Title: Optimal Morphine Dosing Schedule for Neonatal Abstinence Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Anna Thomas, Assistant Professor of Clinical Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1910620136
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Results first posted 2022-09-08 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Neonatal Abstinence Syndrome; Neonatal Opioid Withdrawal; Neonatal Opioid Withdrawal Syndrome
Keywords: morphine; Finnegan
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard (Active Comparator): Infants randomized to the standard arm will receive morphine based on the current institutional treatment protocol: oral morphine 0.05 mg/kg/dose given every 3 hours, initiated if threshold Finnegan score is met. Once stabilized, dose will be weaned by 10% of peak dose per day until discontinuation.
  Interventions: Drug: Morphine scheduled
- Study (Experimental): Infants randomized to the study arm will receive oral morphine 0.05 mg/kg/dose as needed for an elevated Finnegan score. May receive morphine as frequently as every 3 hours if needed.
  Interventions: Drug: Morphine PRN

INTERVENTIONS:
Drug: Morphine PRN — Dose given every 3 hours as-needed for severe NAS, defined by a threshold Finnegan score.
  Other Names: morphine; morphine sulfate
  Arms: Study
Drug: Morphine scheduled — Dose given every 3 hours on a scheduled basis and slowly weaned once stabilized.
  Other Names: morphine; morphine sulfate
  Arms: Standard

SUMMARY:
Randomized pilot trial comparing scheduled morphine dosing with a weaning protocol to intermittent morphine dosing on an as-needed basis for newborns with neonatal abstinence syndrome.

ELIGIBILITY:
Inclusion Criteria:

* newborn greater than or equal to 35 weeks gestation
* intrauterine opioid exposure
* signs and symptoms of opioid withdrawal

Exclusion Criteria:

* congenital anomalies or suspected genetic condition
* co-morbid conditions that require sedation or analgesia due to clinical condition
* ongoing need for respiratory support

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Health Methodist Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard | Study
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard | Study | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Customized [Mean (Standard Deviation); unit: weeks] — Gestational age at birth
  weeks | 37.8 (1.4) | 37.8 (1.8) | 37.8 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 3 | 4 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Buprenorphine exposure [Count of Participants; unit: Participants] | 7 | 3 | 10
Breastfed during hospital stay [Count of Participants; unit: Participants] | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Enrollment Rate
Description: Percentage of eligible subjects who were enrolled and randomized in the study
Time Frame: Prior to second dose of morphine, within 4 hours
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Patients: All eligible patients who were screened for enrollment.
Arm/Group | Eligible Patients
Number analyzed (Participants) | 34
Participants | 17

2. Primary Outcome: Drop Out Rate
Description: Percentage of enrolled subjects who do not complete participation
Time Frame: Through final follow-up call at 6 weeks of age
Measure: Count of Participants; unit: Participants
Groups:
- All Enrolled Subjects: All subjects in each arm.
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 17
Participants | 4

3. Primary Outcome: Number of Study Group Subjects Switched to Standard Arm
Description: Number of study group infants removed from study protocol and treated under standard care.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Study
Number analyzed (Participants) | 8
Participants | 0

4. Secondary Outcome: Length of Hospital Stay From Birth to Discharge
Description: Duration of hospitalization in days
Time Frame: Until discharge, up to 6 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard | Study
Number analyzed (Participants) | 9 | 8
days | 14.6 (4.2) | 11.6 (5.3)

5. Secondary Outcome: Total Cumulative Morphine Exposure
Description: Per kilogram based on birth weight
Time Frame: Until discharge, up to 6 weeks
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Standard | Study
Number analyzed (Participants) | 9 | 8
mg/kg | 3.6 (2.4) | 0.2 (0.2)

6. Secondary Outcome: Peak Morphine Dose
Description: Per kilogram based on birth weight
Time Frame: Until discharge, up to 6 weeks
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Standard | Study
Number analyzed (Participants) | 9 | 8
mg/kg | 0.09 (0.06) | 0.05 (0.02)

7. Secondary Outcome: Length of Morphine Treatment
Description: Duration of morphine treatment in days
Time Frame: Until discharge, up to 6 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard | Study
Number analyzed (Participants) | 9 | 8
days | 11.5 (2.8) | 2.9 (2.3)

ADVERSE EVENTS:
Time Frame: From enrollment to follow-up at 6 weeks post-discharge.
Description: Follow-up adverse events included hospital readmission for withdrawal symptoms, growth failure or failure to thrive. The timing of follow-up at 6 weeks post-discharge varied among participants as it was dependent on length of hospital stay.
Arm/Group | Standard | Study
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 2/9 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard (N=9) | Study (N=8)
over-sedation (Nervous system disorders) | 2 (2) | 0 (0) — Two infants experienced increased somnolence (over-sedation) after escalation of the morphine dose which affected level of alertness and ability to orally feed. This was remedied by decreasing the dose of morphine.

LIMITATIONS AND CAVEATS:
The goal number of subjects was 24 and this was not achieved, which is a limitation. We found that social factors, such as adoption plans and foster placement, limited enrollment of otherwise eligible subjects and resulted in difficulty with follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/53/NCT04298853/Prot_SAP_000.pdf